CLINICAL TRIAL: NCT06080555
Title: A Randomized, Open-label, Parallel, Two-treatment, Single-dose Bioequivalence Study of Ferric Carboxymaltose Injection in Participants With Iron Deficiency Anaemia Under Fasting Conditions
Brief Title: Bioequivalence Study of Ferric Carboxymaltose Injection in Participants With Iron Deficiency Anaemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Collaborators: The First Hospital of Jilin University (Other); Suzhou Guochen Biotek Co., Ltd. (Unknown); Boji Data Technology (Beijing) Co., Ltd. (Unknown); Boji Medical Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023BE-SJMYTT
Record Dates: First submitted 2023-09-27; First posted 2023-10-12 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2023-11

CONDITIONS: Iron Deficiency; Anaemia
Keywords: Bioequivalence
MeSH Terms: conditions — Iron Deficiencies; Anemia | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product-Ferric carboxymaltose Injection provided by SichuanHuiyuPharma (Experimental)
  Interventions: Drug: Ferric Carboxymaltose Injection
- Reference product-marketed by Vifor France (Active Comparator)
  Interventions: Drug: Ferric Carboxymaltose Injection [Ferinject]

INTERVENTIONS:
Drug: Ferric Carboxymaltose Injection — For the T group, participants will have a standardized dinner on the night before the trial, followed by a fasting period of at least 10 h before receiving the test product (T, 10 mL: 500 mg elemental iron) via intravenous injection in the single upper limb, at a continuous rate for 5 min, with a speed of 2 mL/min.
  Arms: Test product-Ferric carboxymaltose Injection provided by SichuanHuiyuPharma
Drug: Ferric Carboxymaltose Injection [Ferinject] — For the R group, participants will have a standardized dinner on the night before the trial, followed by a fasting period of at least 10 h before receiving the reference product (trade name: Ferinject®) (R, 10 mL: 500 mg elemental iron) via intravenous injection on an empty stomach, at a continuous rate for 5 min, with a speed of 2 mL/min.
  Arms: Reference product-marketed by Vifor France

SUMMARY:
The goal of this clinical trial is to compare the pharmacokinetic profile of the developed drug product and reference product in participants with iron deficiency anaemia under fasting condition. The main questions it aims to answer are:

* [Question 1] Is there significant difference in the pharmacokinetic profile between the ferric carboxymaltose injection (10 mL: 500 mg [calculated by iron]) provided by Sichuan Huiyu Pharmaceutical Co., Ltd. and the ferric carboxymaltose injection (trade name: Ferinject®, strength: 10 mL: 500 mg [calculated by iron]) held by Vifor France?
* [Question 2] Is it safe for patient to take ferric carboxymaltose injection (10 mL: 500 mg [calculated by iron]) provided by Sichuan Huiyu Pharmaceutical Co., Ltd. under fasting condition? Participants will be randomly divided into two groups by stratified blocked randomization, with equal number of patients in each group,to receive test product or reference product according to the protocol below.
* Dosing on D1: Group T (Test product) Group R (Reference product)
* PK blood sample collection
* Safety evaluation

ELIGIBILITY:
Inclusion Criteria:(all inclusion criteria must be met to be included)

1. Participants with a thorough understanding of the content, process, and potential adverse reactions of the study, who have signed Informed Consent Form;
2. Those able to complete the study as per the study protocol;
3. Participants (including their partners) having no planning for pregnancy from the screening through 3 months after the last administration, and willing to take effective contraceptive measures;
4. Male and/or female participants aged 18-60 (including those aged 18 and 60);
5. Male participants weighing not less than 50 kilograms and female participants weighing not less than 45 kilograms. Body mass index (BMI) = weight (kg)/height 2 (m2), with a body mass index ranging from 18 to 30 kg/m2 (including both boundaries);
6. Diagnosis of iron-deficiency anemia is confirmed during the screening process based on the following criteria (both criteria must be met): ①Hemoglobin (Hb) < 110 g/L (for females) or Hb < 120 g/L (for males). ②Serum ferritin ≤ 100 ng/mL, or when the serum transferrin saturation (TSAT) is ≤ 30%, serum ferritin ≤ 300 ng/mL.

Exclusion Criteria: (meeting any one of these criteria will result in exclusion)

1. Participants with an allergic constitution, such as asthma and eczema, or having known hypersensitivity to iron, maltose or its analogues, metabolites;
2. In addition to iron-deficiency anemia, participants will be excluded from the screening process if they have had any of the following conditions within the past 6 months: cardiovascular, digestive, respiratory, urinary, hematological, metabolic, immune, or neurological system diseases, or any active malignancies as determined by the investigator;
3. Individuals with acute infection in previous 2 weeks prior to the screening visit;
4. laboratory tests: alanine aminotransferase (ALT) > 1.5 times the upper limit of the normal range (× ULN); aspartate transaminase (AST) > 1.5 × ULN; total serum bilirubin (TBiL) > 1.5 × ULN; albumin < 30 g/L; platelet count < 90 × 109/L; neutrophil absolute count < 1.3 × 109/L; glomerular filtration rate < 60 mL/min/1.73 m2 (estimated based on simplified Modification of Diet in Renal Disease (MDRD) formula);
5. Serious arrhythmias showed in ECG at screening period, such as recurrent and highly symptomatic ventricular tachycardia, atrial fibrillation accompanied by rapid ventricular response or supraventricular tachycardia, and are not suitable for the trial at the investigator's discretion;
6. With history of iron storage diseases such as haemochromatosis; history of iron utilisation disorders such as sideroachrestic anaemia; history of haemoglobinopathy (such as Thalassemia); having symptomatic anemia requiring red blood cell infusion;
7. Receiving IV iron therapy in previous 3 months prior to the screening visit, erythropoiesis stimulating agent (ESA) therapy and/or blood transfusion in previous 4 weeks prior to the screening visit, and oral iron or iron-containing products in previous 7 days prior to the screening visit;
8. Receiving any prescription drugs that affect PK results in previous 14 days prior to the screening visit;
9. Receiving any non-prescription drugs, traditional Chinese medicine, or healthcare products that affect PK results in previous 7 days prior to the screening visit;
10. Individuals who consume an average of more than 5 cigarettes per day in previous 3 months prior to the screening visit;
11. Individuals who have undergone surgeries within the past 3 months that might affect drug absorption, distribution, metabolism, or excretion, or those who are planning to undergo surgeries during the study period, will also be deemed ineligible to participate;
12. Received investigational drug or participated in other clinical trials within the preceding 3 months;
13. Blood donation or significant blood loss in previous 3 months prior to the screening visit (> 400 mL, excluding menstrual blood loss in female participants);
14. Female participants who are currently breastfeeding or have positive pregnancy test results during the screening period or clinical trials;
15. People having viral hepatitis, such as hepatitis B or C, HIV antibody positive, treponema pallidum antibody positive and rapid plasma reaction (RPR) positive; (patients with positive hepatitis B surface antigen alone can be subjected to additional test for HBV DNA, patients with positive hepatitis C antibody alone can be subjected to additional test for HCV RNA, and those with positive Treponema pallidum antibody alone can be subjected to additional test for RPR);
16. Individuals with a history of drug abuse in previous 5 years prior to the screening visit or those who have used drugs in previous 3 months prior to the screening visit;
17. Acute illness or concomitant medication from the screening stage to the study drug dosing;
18. Having chocolate, or any food or drink containing caffeine or rich in xanthine 48 h before receiving the study drug;
19. Regular drinkers in previous 3 months prior to the screening visit, i.e. those who consume an average of over 2 units of alcohol per day (1 unit = 360 mL of beer or 45 mL of 40% liquor or 150 mL of wine), or those who are unwilling to give up drinking or any alcoholic products during the trial period;
20. Those with positive drug abuse screening or alcohol screening;
21. Having special diet, such as grapefruit or products containing grapefruit ingredients, taking strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, and excretion, within 48 h before receiving the study drug;
22. Those receiving non-inactivated vaccine in previous 14 days prior to the screening visit or planning to receive vaccine during the study period;
23. Those who cannot tolerate venipuncture or have a history of fear of needles or hemophobia;
24. Other circumstances that may increase the risk of the participant or interfere with the evaluation or results of the study at the investigator's discretion;
25. Participants not suitable for the trial at the investigator's discretion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of total iron in serum: Cmax | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  Cmax is the peak concentration of total iron in serum. It is directly obtained from observed blood drug concentration-time data.
Pharmacokinetic parameter of total iron in serum: AUC0-t | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  AUC0-t is the area under the concentration curve from dosing to the last measurable blood drug concentration.It is calculated using the linear trapezoidal rule.
Pharmacokinetic parameter of transferrin bound iron in serum: Cmax | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  Cmax is the peak concentration of transferrin bound iron in serum. It is directly obtained from observed blood drug concentration-time data.
Pharmacokinetic parameter of transferrin bound iron in serum: AUC0-t | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  AUC0-t is the area under the concentration curve from dosing to the last measurable blood drug concentration.It is calculated using the linear trapezoidal rule.

SECONDARY OUTCOMES:
Pharmacokinetic parameter of total iron in serum: AUC0-∞ | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  AUC0-∞ is the area under the curve from dosing to extrapolated infinite time. AUC0-∞ = AUC0-t + Ct / λz, where Ct is the last measurable concentration, and λz is the elimination rate constant.
Pharmacokinetic parameter of total iron in serum: Tmax | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  Tmax is the time to reach maximum concentration of total serum iron.
Pharmacokinetic parameter of total iron in serum: t1/2 | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  t1/2 is the terminal elimination half-life of total serum iron. It is calculated as ln2 / λz.
Pharmacokinetic parameter of total iron in serum:λz | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  λz is the elimination rate constant of total serum iron. It is calculated as the negative reciprocal of the slope of the terminal phase of the logarithm-linear drug concentration-time curve using linear regression.
Pharmacokinetic parameter of transferrin bound iron in serum: AUC0-∞ | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  AUC0-∞ is the area under the curve from dosing to extrapolated infinite time. AUC0-∞ = AUC0-t + Ct / λz, where Ct is the last measurable concentration, and λz is the elimination rate constant.
Pharmacokinetic parameter of transferrin bound iron in serum: Tmax | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  Tmax is the time to reach maximum concentration of serum transferrin bound iron.
Pharmacokinetic parameter of transferrin bound iron in serum: t1/2 | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  t1/2 is the terminal elimination half-life of transferrin bound iron. It is calculated as ln2 / λz.
Pharmacokinetic parameter of transferrin bound iron in serum:λz | 24hours,12hours,0hour before administration, and 5minutes,10minutes,15minutes,30minutes,45minutes,1hour,1.5hours,2hours,4hours,6hours,8hours,10hours,12hours,24hours,36hours,48hours,72hours,96hours,120hours and 144hours after administration.
  λz is the elimination rate constant of transferrin bound iron. It is calculated as the negative reciprocal of the slope of the terminal phase of the logarithm-linear drug concentration-time curve using linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Li Xiang, Study Director — Sichuan Huiyu Pharmaceutical Co., Ltd
Locations (4):
- China (4):
  - Boji medical technology (Beijing) co., Ltd, Beijing, Beijing Municipality
  - Boji Medical Technology Co., Ltd, Guangzhou, Guangdong
  - Suzhou Guochen Biotek Co., Ltd, Suzhou, Jiangsu
  - Phase I Clinical Trial Department, The First Hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ikuta K, Shimura A, Terauchi M, Yoshii K, Kawabata Y. Pharmacokinetics, pharmacodynamics, safety, and tolerability of intravenous ferric carboxymaltose: a dose-escalation study in Japanese volunteers with iron-deficiency anemia. Int J Hematol. 2018 May;107(5):519-527. doi: 10.1007/s12185-018-2400-z. Epub 2018 Jan 22. PMID 29357079
- [Background] Ding Y, Zhu X, Li X, Zhang H, Wu M, Liu J, Palmen M, Roubert B, Li C. Pharmacokinetic, Pharmacodynamic, and Safety Profiles of Ferric Carboxymaltose in Chinese Patients with Iron-deficiency Anemia. Clin Ther. 2020 Feb;42(2):276-285. doi: 10.1016/j.clinthera.2019.12.010. Epub 2020 Jan 11. PMID 31937462
- [Background] Ferric Carboxymaltose Injection Package Insert. Vifor (International) Inc
- [Background] Multidisciplinary Expert Consensus on Diagnosis, Treatment, and Prevention of Iron Deficiency and Iron-Deficiency Anemia by the Hematology Branch of the Chinese Medical Association (Anemia Group) [J]. Chinese Medical Journal, 2022, 102(41):3246-3256
- See also: EMA Guideline on the investigation of bioequivalence — https://www.ema.europa.eu/en/documents/scientific-guideline/guideline-investigation-bioequivalence-rev1_en.pdf
- See also: EMA Reflection paper on the data requirements for intravenous iron-based nano-colloidal products developed with reference to an innovator medicinal product — https://www.ema.europa.eu/en/documents/scientific-guideline/reflection-paper-data-requirements-intravenous-iron-based-nano-colloidal-products-developed_en.pdf